CLINICAL TRIAL: NCT00061620
Title: Phase I Study of Continuous Infusion Schedule of (E)-2'-Deoxy-2'-(Fluoromethylene) Cytidine (Tezacitabine, FMdC) in Hematologic Malignancies
Brief Title: Phase I Study of Continuous Infusion Schedule of FMdC in Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Chiron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-168
Record Dates: First submitted 2003-05-30; First posted 2003-06-02 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Hematologic Malignancies
Keywords: Investigational; Chemotherapy; Hematologic Malignancies; Nucleoside analogue
MeSH Terms: conditions — Hematologic Neoplasms | interventions — tezacitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tezacitabine (Experimental): Tezacitabine as a bolus infusion daily x 5
  Interventions: Drug: Tezacitabine (FMdC)

INTERVENTIONS:
Drug: Tezacitabine (FMdC) — 7.5 mg/m2 bolus infusion daily x 5
  Other Names: FMdC; (E)-2'-Deoxy-2'-(Fluoromethylene) Cytidine

SUMMARY:
The goal of this clinical research study is to find the highest dose of Tezacitabine (FMdC) which can be safely given as a continuous infusion by vein to patients with hematologic malignancies. The general safety and effectiveness of this drug will also be studied.

DETAILED DESCRIPTION:
Patients with leukemias that have relapsed from previous therapies have a low cure rate. Hence the need to discover new antileukemic agents. Tezacitabine is a nucleoside analogue with equivalent or even superior activity when compared with ara-C in leukemic cell lines. It has shown significant antitumor activity in vitro and in vivo tumor models. Several phase I studies with various dosing schedules have been conducted in solid tumors where the dose-limiting toxicity (DLT) is mainly myelosuppression, usually a favorable feature for development of leukemia. In a phase I study in hematological malignancies, we used Tezacitabine as a bolus infusion daily x 5. The DLT consisted of grade 3 CNS toxicities and mucositis in 3/6 patients. The study is ongoing and we are currently evaluating a dose level of 7.5 mg/m2 as possible Maximum Tolerated Dose (MTD). However, in view of the fact that tezacitabine is a cell cycle specific agent with a short terminal plasma half-life of 2 to 6 hours, a continuous infusion dosing schedule may enhance the activity and reduce the incidence of adverse effects of tezacitabine.

ELIGIBILITY:
* Patient with relapsed/refractory acute leukemias (AML, ALL, high-grade myelodysplastic syndromes, CMML in transformation with >/= 10% peripheral blood/bone marrow blasts, CML in blast crisis), or patients with relapsed/refractory CLL and an absolute neutrophil count of >/= 1,000/ml and platelet count of >/= 75,000/ml.
* Signed informed consent indicating that patients are aware of the investigational nature of this study, and in keeping with the policies of this hospital. The only acceptable consent form is attached at the end of this protocol.
* Age >/= 15 years.
* ECOG performance status </= 2.
* No severe, concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for study entry.
* Pregnant and/or lactating females are not eligible.
* Normal organ function (serum bilirubin £ 2 mg/dL, serum creatinine £ 2 mg/dL). Patients with renal or liver dysfunction due to organ leukemic involvement may be eligible after discussion with the principle investigator.
* Patients must be off of all previous chemotherapy, immunotherapy, or radiotherapy for at least 2 weeks prior to entering this study, and must have recovered from all toxic effects, unless life-threatening increases in tumor burden occur.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-09-06 (Actual); Primary Completion 2004-02-12 (Actual); Study Completion 2004-02-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD)
  MTD determination made from dose level without a dose-limiting toxicity (DLT)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Faderl, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center's website — http://www.mdanderson.org